CLINICAL TRIAL: NCT02012985
Title: A Phase 1/2, Randomised, Placebo-controlled, Double-blind, Multi-centre Study to Evaluate the Efficacy and Safety of OC5 to Reduce Urinary Oxalate in Subjects With Primary Hyperoxaluria
Brief Title: Study to Evaluate the Efficacy and Safety of Oxabact (OC5) in Patients With Primary Hyperoxaluria
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: OxThera (Industry)
Collaborators: FP7-SME-2013 Research for the benefit of SMEs program (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OC5-DB-01
Record Dates: First submitted 2013-12-11; First posted 2013-12-17 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Primary Hyperoxaluria
Keywords: hyperoxaluria; oxalate; PH
MeSH Terms: conditions — Hyperoxaluria, Primary; Hyperoxaluria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxabact OC5 capsules (Experimental): The active study drug consists of Oxalobacter formigenes OC5 in enteric-coated size-4 capsules. The dose (not less than (NLT) 1E+09 colony forming units (CFU)) will be administrated orally with breakfast and dinner as one capsule two times per day for 8 to 10 weeks.
  Interventions: Biological: Oxabact OC5 capsules
- Placebo capsules (Placebo Comparator): The placebo study drug consists of microcrystalline cellulose in enteric-coated size-4 capsules. It has been manufactured to mimic the OC5 capsule. The dose will be administrated orally with breakfast and dinner as one capsule two times per day for 8 to 10 weeks.
  Interventions: Drug: Placebo capsules

INTERVENTIONS:
Biological: Oxabact OC5 capsules — The dose will be not less than (NLT) 1E+09 colony forming units (CFU) twice daily for 8 to 10 weeks. The dose (an enteric-coated size 4 capsule) will be administered orally with breakfast and dinner.
  Other Names: Oxalobacter formigenes
  Arms: Oxabact OC5 capsules
Drug: Placebo capsules — An enteric-coated placebo capsule manufactured to mimic the OC5 capsule. The capsule will be administered orally with breakfast and dinner twice daily for 8 to 10 weeks.
  Arms: Placebo capsules

SUMMARY:
The purpose of this study is to determine if Oxalobacter formigenes is effective at lowering urinary oxalate levels in patients with primary hyperoxaluria.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent (as applicable for the age of the subject).
* Male or female subjects ≥ 2 years of age (Germany & France) / Male or female subjects ≥ 5 years of age (United Kingdom)
* A diagnosis of PH type I, II or III (as determined by standard diagnostic methods).
* A mean urinary oxalate excretion of > 1.0 mmol/24h/1.73m2, based on at least three eligible urine collections performed during baseline (weeks 1-4).
* Renal function defined as an estimated GFR ≥ 40 ml/min normalised to 1.73m2 body surface area, or a creatinine clearance of ≥ 40 ml/min normalised to 1.73m2 body surface area.
* Subjects receiving vitamin B6 must be receiving a stable dose for at least 3 months prior to screening and must not change the dose during the study. Subjects not receiving vitamin B6 at study entry must be willing to refrain from initiating pyridoxine during study participation.

Exclusion Criteria:

* Inability to collect complete 24-hour urine samples. Each urine collection will be evaluated for completeness based on urine qualitative criteria.
* Inability to swallow size 4 capsules twice daily for 8 to 10 weeks.
* Subjects that have undergone transplantation (solid organ or bone marrow).
* The existence of secondary hyperoxaluria, e.g. hyperoxaluria due to bariatric surgery or chronic gastrointestinal diseases such as cystic fibrosis, chronic inflammatory bowel disease and short-bowel syndrome.
* Use of antibiotics to which O. formigenes is sensitive, including chronic use, a history of more than two courses of antibiotic use during the past 6 months, current antibiotic use, or antibiotics use within 14 days of initiating study medication.
* Subjects who require immune suppressive therapy.
* Current treatment with ascorbic acid preparation.
* Pregnancy.
* Women of child-bearing potential who are not using adequate contraceptive precautions such as oral, transdermal, injectable, or implanted contraceptives, IUD, complete abstinence, use of a condom by the sexual partner, or sterile sexual partner.
* Presence of a medical condition that the Principal Investigator considers likely to make the subject susceptible to adverse effect of study treatment or unable to follow study procedures.
* Participation in any study of an investigational product, biologic, device, or other agent within 30 days prior to screening or not willing to forego other forms of investigational treatment during this study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in urinary oxalate levels from Baseline to week 8 of treatment. | 8 weeks of active treatment (i.e. between Weeks 7 and 14 of the study)

SECONDARY OUTCOMES:
Change in urinary oxalate levels from Baseline to week 8 of treatment in subsets of subjects | 8 weeks of active treatment (i.e. between Weeks 7 and 14 of the study)
  Change in urinary oxalate levels from Baseline to week 8 of treatment in subsets of subjects defined by:
  * baseline urinary oxalate level, above and below 1.5 mmol/24h/1.73m2
  * concomitant vitamin B6 therapy and no vitamin B6 therapy
  * eGFR of ≥90 mL/min/1.73m2 (normal renal function) and < 90 mL/min/1.73m2 (mild to moderate reduction in renal function)
  * age below 18 and age 18 or above
Number of subjects who reach urinary oxalate levels below 0.5, 0.7 and 1.0 mmol/24h/1.73m2 respectively from Baseline to week 8 of treatment. | 8 weeks of active treatment (i.e. between Weeks 7 and 14 of the study)
Change in plasma oxalate levels from Baseline to week 8 of treatment. | 8 weeks of active treatment (i.e. between Weeks 7 and 14 of the study)
Change in urinary oxalate levels from Baseline to week 4 of treatment. | 8 weeks of active treatment (i.e. between Weeks 7 and 10 of the study)
Correlation between change in plasma oxalate levels and change in urinary oxalate levels, from Baseline to week 8 of treatment. | 8 weeks of active treatment (i.e. between Weeks 7 and 14 of the study)
Change in number of O. formigenes in faeces from Baseline to week 8 of treatment. | 8 weeks of active treatment (i.e. between Weeks 7 and 14 of the study)
Adverse events | 8 weeks of active treatment (i.e. between Weeks 7 and 14 of the study)
Haematology | 14 weeks (Throughout the study)
  Blood samples taken for hematology at weeks 0, 5, 10 and 14. Complete blood count with differential and platelet count evaluated.
Clinical Chemistry | 14 weeks (Throughout the study)
  Blood samples taken for clinical chemistry at weeks 0, 5, 10 and 14. Blood Urea Nitrogen, creatinine, electrolytes (Na+, K+, Mg++, Ca++, HCO3+, Cl), glucose, pH, albumin, alkaline phosphatase, ALT, AST, total bilirubin and total protein evaluated.
Urinalysis | 14 weeks (Throughout the study)
  Urine samples will be taken at weeks 0, 5, 10 and 14 of the study. Protein, glucose and pH evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Hoppe, MD PhD, Principal Investigator — Universitätsklinikum Bonn, Dept of Paediatric Nephrology
Locations (8):
- France (4):
  - Hôpital Robert-Debré, Néphrologie Pédiatrique, Paris, Cedex 19
  - Hôpital des Enfants, Centre de référence maladies rénales rares du Sud-Ouest (SORARE), CHU de Bordeaux, Bordeaux
  - Hôpital Femme Mère Enfant, Lyon - Paediatric Dept, Lyon
  - Hôpital Necker-Enfants Malades,Centre de référence des Maladies Rénales Héréditaires de l'Enfant et de l'Adulte (MARHEA), Paris
- Universitätsklinikum Bonn, Dept of Paediatric Nephrology, Bonn, Germany
- United Kingdom (3):
  - Birmingham Children's Hospital NHS Foundation Trust - Dept of Nephrology, Birmingham
  - Royal Free Hospital -UCL Centre for Nephrology, London
  - Great Ormond Street Hospital for Children NHS Trust, London